CLINICAL TRIAL: NCT00888654
Title: Phase II Trial of B-DIM (DIM: 3,3 Diindolylmethane) on Intermediate Endpoint Biomarkers in Patients With Prostate Cancer Who Are Undergoing Prostatectomy
Brief Title: Diindolylmethane in Treating Patients With Stage I or Stage II Prostate Cancer Undergoing Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000641168; P30CA022453 (NIH); WSU-2007-128
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- B-Dim, Radical Prosatectomy (Experimental): B-DIM 225 mg orally twice daily x 14-72 days (based on scheduling of surgery)
  Radical Prostatectomy
  Interventions: Drug: B-Dim; Procedure: Radical Prosatectomy

INTERVENTIONS:
Drug: B-Dim — B-DIM 225 mg orally twice daily x 14-72 days (based on scheduling of surgery)
  Other Names: 3,3'-Diindolylmethane
Procedure: Radical Prosatectomy
  Other Names: therapeutic conventional surgery

SUMMARY:
RATIONALE: The use of diindolylmethane, a substance found in cruciferous vegetables, may slow the growth of tumor cells.

PURPOSE: This phase II trial is studying how well diindolylmethane works in treating patients with stage I or stage II prostate cancer undergoing radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure the level of diindolylmethane in prostate tissue after treatment with oral microencapsulated diindolylmethane (B-DIM) in patients with stage I or II adenocarcinoma of the prostate undergoing radical prostatectomy.

Secondary

* To measure serum biomarkers (e.g., total PSA, serum testosterone, and diindolylmethane levels) pre- and post-treatment with B-DIM.
* To measure tissue biomarkers (e.g., androgen receptor, NF-κB, and PSA) pre- and post-treatment with B-DIM.

OUTLINE: This is a multicenter study.

Patients receive oral microencapsulated diindolylmethane (B-DIM) twice daily for 14-72 days in the absence of disease progression or unacceptable toxicity. Patients then undergo radical prostatectomy 1 day after the last dose of B-DIM.

Patients undergo blood and tissue sample collection for correlative laboratory studies. Blood samples are analyzed for serum PSA, testosterone, and diindolylmethane levels by high performance liquid chromatography and tandem mass spectrometry (LC-MS/MS). Tissue samples are analyzed for diindolylmethane concentration by LC-MS/MS and for androgen receptor, activated NF-κB (p65 antibody), and PSA expression by IHC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Stage I or II (T1-T2 a, b, or c) disease
  * Disease confined to the prostate by clinical judgment of the surgeon
* Deemed an appropriate candidate for surgery by clinical judgment of the surgeon

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and/or ALT ≤ 2.5 times ULN if alkaline phosphatase normal OR alkaline phosphatase ≤ 4 times ULN if AST and/or ALT normal
* Serum creatinine ≤ 2.0 mg/dL
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to oral microencapsulated diindolylmethane
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive hart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, hormonal therapy, brachytherapy, cryotherapy, external beam radiotherapy, or other therapy for prostate cancer
* No concurrent micronutrient supplements or dietary soy products
* No concurrent systemic therapy for any other cancer
* No concurrent p450 inducers or inhibitors (e.g., carbamazepine, clarithromycin, fluconazole, fosphenytoin, itraconazole, ketoconazole, phenobarbital, phenytoin, rifabutin, or rifampin)
* No concurrent finasteride or dutasteride
* No other concurrent investigational or commercial agents or therapies for the malignancy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth I. Heath, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- B-Dim, Radical Prosatectomy: B-DIM 225 mg orally twice daily x 14-72 days (based on scheduling of surgery)
  Radical Prostatectomy
  B-Dim: B-DIM 225 mg orally twice daily x 14-72 days (based on scheduling of surgery)
  Radical Prosatectomy
Period: Overall Study
Arm/Group | B-Dim, Radical Prosatectomy
Started | 41
Completed | 31
Not Completed | 10
Not completed — Problems swallowing oral meds. | 1
Not completed — Not enough oral meds before surgery | 3
Not completed — Surgery aborted | 2
Not completed — Withdrawal by Subject | 1
Not completed — Inelig. due to contraindication of med | 1
Not completed — Change in surg date | 1
Not completed — Stopped meds due to headaches | 1

BASELINE CHARACTERISTICS:
Arm/Group | B-Dim, Radical Prosatectomy
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 58 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Mean Level of Diindolylmethane in Prostate Tissue After Treatment
Time Frame: Within the first 24 months after radical prostatectomy.
Population: Patients that were eligible, evaluable, and compliant
Measure: Mean (90% Confidence Interval); unit: ng/g
Arm/Group | B-Dim, Radical Prosatectomy
Number analyzed (Participants) | 28
ng/g | 14.2 [10.6 to 17.7]

2. Secondary Outcome: Serum Levels of PSA, Testosterone, and Diindolylmethane
Description: Serum levels of PSA, testosterone, and diindolylmethane (DIM)
Time Frame: Pre and post radical prostatectomy
Population: All enrolled patients except for one patient who was deemed ineligible due to a disallowed concomitant medication and for one patient whose prostatectomy was cancelled because of adhesions found at the time of surgery.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | B-Dim, Radical Prosatectomy
Number analyzed (Participants) | 39
ng/ml
  Pre-treatment PSA | 6.4 [2.1 to 29.4]
  Post-treatment PSA | 5.8 [2.6 to 28.3]
  Pre-treatment Testosterone | 301 [77 to 608]
  Post-treatment Testosterone | 388 [110 to 686]
  Pre-treatment DIM | 0.0 [0.0 to 0.0]
  Post-treatment DIM | 7.5 [0.0 to 24.7]

3. Secondary Outcome: Levels of Androgen Receptor in Prostate Tissue
Description: Levels of androgen receptor in prostate tissue as measured by AR score (intensity x % cells stained), higher scores indicate higher levels of androgen receptor in prostate tissue.
Time Frame: Pre and post radical prostatectomy
Population: as for outcome 2
Measure: Mean (90% Confidence Interval); unit: AR score (intensity x % cells stained)
Arm/Group | B-Dim, Radical Prosatectomy
Number analyzed (Participants) | 39
AR score (intensity x % cells stained)
  Pre-BR-DIM Androgen Receptor | 278 [263 to 293]
  Post-BR-DIM Androgen Receptor | 245 [227 to 263]

ADVERSE EVENTS:
Arm/Group | B-Dim, Radical Prosatectomy
Serious Adverse Events (participants affected / at risk) | 2/41
Other Adverse Events (participants affected / at risk) | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-Dim, Radical Prosatectomy (N=41)
Headache (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
There were no significant limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes